CLINICAL TRIAL: NCT04416763
Title: Diagnostic Value of Endoscopic Ultrasound Elastography and Contrast Enhanced Endoscopic Ultrasound for Differential Diagnosis of Gallbladder Polyp
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Other Study IDs: H-2005-135-1124
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Gallbladder Polyps or Masses Greater Than 8-10 mm in Size
Keywords: Gallbladder polyp; Endoscopic ultrasound; Elastography; contrast enhanced endoscopic ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gallbladder polyps are often detected incidentally by ultrasonography. The most of gallbladder polyps are non-neoplastic such as cholesterol polyps and do not need further treatments. However, neoplastic polyps, which need additional treatments to prevent malignancy, show the same appearance on ultrasound. Clinically, the differential diagnosis between cholesterol polyps and adenomatous polyps is very important for patient follow-up and treatment. However, differential diagnosis between these two conditions is difficult using conventional trans-abdominal ultrasound.

Endoscopic ultrasound (EUS) is less affected and disturbed by subcutaneous fat or intraabdominal air, so a clearer image of pancreatobiliary system can be obtained. In addition, EUS elastography and contrast enhanced EUS are recently introduced. EUS elastography enables practitioners to evaluate the stiffness of a target lesion and compare it with surrounding tissues (strain ratio). Also, contrast enhanced EUS is used widely with additional information such as presence of vessels and enhancement pattern of soft tissues. Several studies have been published that EUS elastography can help in the differential diagnosis of pancreatic solid lesions.

Although studies have been conducted to confirm the usefulness of transabdomnial ultrasound with elastography or contrast enhancement at differentiating gallbladder polyps, no prospective studies have been conducted to evaluate the usefulness of EUS elastography or contrast enhanced EUS for gallbladder polyp. Therefore, with this prospective study, we would like to evaluate the diagnostic value of EUS elastography and contrast enhanced EUS for differential diagnosis of gallbladder polyps.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Gallbladder polyp of 8-10mm or more in size confirmed by imaging tests
   2. Must be 19 years old or older
   3. With voluntary agreement to participate in the study after be informed about the necessity of EUS due to the clinical necessity
2. Exclusion Criteria:

   1. Unable to confirm histological diagnosis (ex. Patients did not underwent cholecystectomy)
   2. Younger than 18 year-old
   3. Without agreement with this study or informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have GB polyps and are recommended cholecystectomy due to large size of polyp (8-10 mm or larger).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Pathologic diagnosis of gallbladder polyp after cholecystectomy | within 10 days after operation
  Pathologic diagnosis of gallbladder polyps or masses in cholecystectomy specimen
Difference of strain ratio | Within two years of starting the study
  Differences in strain ratio between non-neoplastic and neoplastic gallbladder polyps.

SECONDARY OUTCOMES:
Optimal cut-off valve of strain ratio | Within two years of starting the study
  Optimal cut-off valve of strain ratio for differential diagnosis between cholesterol polyps and adenomatous polyps
Diagnostic value of EUS-elastography | Within two years of starting the study
  Sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy of EUS-elastography for diagnosis of cholesterol polyps.
Diagnostic value of contrast enhanced EUS | Within two years of starting the study
  Sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy of contrast enhanced EUS for diagnosis of cholesterol polyps.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Corwin MT, Siewert B, Sheiman RG, Kane RA. Incidentally detected gallbladder polyps: is follow-up necessary?--Long-term clinical and US analysis of 346 patients. Radiology. 2011 Jan;258(1):277-82. doi: 10.1148/radiol.10100273. Epub 2010 Aug 9. PMID 20697115
- [Background] Park CH, Chung MJ, Oh TG, Park JY, Bang S, Park SW, Kim H, Hwang HK, Lee WJ, Song SY. Differential diagnosis between gallbladder adenomas and cholesterol polyps on contrast-enhanced harmonic endoscopic ultrasonography. Surg Endosc. 2013 Apr;27(4):1414-21. doi: 10.1007/s00464-012-2620-x. Epub 2012 Dec 12. PMID 23233003
- [Background] Kozuka S, Tsubone N, Yasui A, Hachisuka K. Relation of adenoma to carcinoma in the gallbladder. Cancer. 1982 Nov 15;50(10):2226-34. doi: 10.1002/1097-0142(19821115)50:103.0.co;2-3. PMID 7127263
- [Background] Sugiyama M, Atomi Y, Kuroda A, Muto T, Wada N. Large cholesterol polyps of the gallbladder: diagnosis by means of US and endoscopic US. Radiology. 1995 Aug;196(2):493-7. doi: 10.1148/radiology.196.2.7617866.
- [Background] Choi WB, Lee SK, Kim MH, Seo DW, Kim HJ, Kim DI, Park ET, Yoo KS, Lim BC, Myung SJ, Park HJ, Min YI. A new strategy to predict the neoplastic polyps of the gallbladder based on a scoring system using EUS. Gastrointest Endosc. 2000 Sep;52(3):372-9. doi: 10.1067/mge.2000.108041. PMID 10968853
- [Background] Practical Guidelines for Management of Gallbladder Polyps. Korean Journal of HBP Surgery Vol. 14, No. 3, September 2010
- [Background] Wiles R, Thoeni RF, Barbu ST, Vashist YK, Rafaelsen SR, Dewhurst C, Arvanitakis M, Lahaye M, Soltes M, Perinel J, Roberts SA. Management and follow-up of gallbladder polyps : Joint guidelines between the European Society of Gastrointestinal and Abdominal Radiology (ESGAR), European Association for Endoscopic Surgery and other Interventional Techniques (EAES), International Society of Digestive Surgery - European Federation (EFISDS) and European Society of Gastrointestinal Endoscopy (ESGE). Eur Radiol. 2017 Sep;27(9):3856-3866. doi: 10.1007/s00330-017-4742-y. Epub 2017 Feb 9. PMID 28185005
- [Background] Teber MA, Tan S, Donmez U, Ipek A, Ucar AE, Yildirim H, Aslan A, Arslan H. The use of real-time elastography in the assessment of gallbladder polyps: preliminary observations. Med Ultrason. 2014 Dec;16(4):304-8. doi: 10.11152/mu.201.3.2066.164.1mat. PMID 25463882
- [Background] Kitano M, Kudo M, Sakamoto H, Komaki T. Endoscopic ultrasonography and contrast-enhanced endoscopic ultrasonography. Pancreatology. 2011;11 Suppl 2:28-33. doi: 10.1159/000323493. Epub 2011 Apr 5. PMID 21464584
- [Derived] Cho IR, Lee SH, Choi JH, Chun JW, Lee MW, Lee MH, Kim J, Lee TS, Paik WH, Ryu JK, Kim YT. Diagnostic performance of EUS-guided elastography for differential diagnosis of gallbladder polyp. Gastrointest Endosc. 2024 Sep;100(3):449-456.e1. doi: 10.1016/j.gie.2024.02.015. Epub 2024 Feb 29. PMID 38431102